CLINICAL TRIAL: NCT02813629
Title: Transcranial Direct Current Stimulation Associated With Peripheral Electrical Stimulation for Pain Control in Individuals With Sickle Cell Disease
Brief Title: tDCS Associated With Peripheral Electrical Stimulation for Pain Control in Individuals With Sickle Cell Disease
Acronym: tDCS/PES_SCD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Faculdade Adventista da Bahia (Other)
Collaborators: Federal University of Bahia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 31237514.1.0000.0042
Record Dates: First submitted 2016-05-10; First posted 2016-06-27 (Estimated); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Anemia, Sickle Cell; Chronic Pain
Keywords: transcranial Direct Current Stimulation; Peripheral Electrical Stimulation; Sickle Cell Disease; Transcutaneous Electrical Nerve Stimulation; quantitative Electroencephalography
MeSH Terms: conditions — Anemia, Sickle Cell; Chronic Pain | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- SS-tDCS (active) plus PES (active) (Active Comparator): tDCS plus PES (n=15).
  Interventions: Device: tDCS plus PES
- SS-tDCS (active) plus PES (simulated) (Active Comparator): tDCS plus PES (n=15).
  Interventions: Device: tDCS plus PES
- SS-tDCS (simulated) plus PES (active) (Active Comparator): tDCS plus PES (n=15).
  Interventions: Device: tDCS plus PES
- SS-tDCS (simulated) plus PES (simulated) (Sham Comparator): tDCS plus PES (n=15).
  Interventions: Device: tDCS plus PES
- SC-tDCS (active) plus PES (active) (Active Comparator): tDCS plus PES (n=15).
  Interventions: Device: tDCS plus PES
- SC-tDCS (active) plus PES (simulated) (Active Comparator): tDCS plus PES (n=15).
  Interventions: Device: tDCS plus PES
- SC-tDCS (simulated) plus PES (active) (Active Comparator): tDCS plus PES (n=15).
  Interventions: Device: tDCS plus PES
- SC-tDCS (simulated) plus PES (simulated) (Sham Comparator): tDCS plus PES (n=15).
  Interventions: Device: tDCS plus PES

INTERVENTIONS:
Device: tDCS plus PES — transcranial direct current stimulation (tDCS) uses a pair of electrodes and sponges soaked in saline solution placed over specific regions of the head to polarize neurons and produce changes in resting membrane potentials. This changes may increase or decrease neuronal excitability and produce diverse clinical effects, including analgesia.
  PES uses also a pair of electrodes over specific regions of the body to promote neuronal action potentials in peripheral nerves. PES over motor threshold increases cortical excitability, and at the sensory threshold decreases excitability.
  Other Names: transcranial direct current stimulation (tDCS); peripheral electrical stimulation (PES)

SUMMARY:
So far, no study investigated the safety and efficacy analgesic of transcranial direct current stimulation (tDCS) associated to peripheral electrical stimulation (PES) in individuals with SCD who suffer from chronic pain. Several studies have reported a decrease in O²Hb concentration in the regions below the electrodes and in other cortical areas during anodic or cathodic tDCS, which implies a risk factor for vasoocclusive events in individuals with SDC due to polymerization of hemoglobin when exposed to these low O²Hb concentrations. For this reasion, the aim main of this study is to assess the effect of a single session of transcranial direct current stimulation (tDCS) associated to peripheral electrical stimulation (PES) on safety and efficacy analgesic in individuals with sickle cell disease (SCD). Others aims sencondaries are evaluate the effect of a single session of transcranial direct current stimulation (tDCS) associated to peripheral electrical stimulation (PES) on biomarkers neurophysiological and inflammatory.

DETAILED DESCRIPTION:
Pain, in its various manifestations, is the symptom most often associated to SCD, being responsible for over 90% of hospital admissions. Oftenly pain has a major impact on the patient's life and is associated with some degree of disability. Chronic pain may reflect the continuity of tissue injury and central nervous system maladaptive plasticity. They start with tissue injuries such as leg ulcers, avascular osteonecrosis, chronic osteomyelitis, arthropathy, or even continue after the repair process, by central nervous sensitization and / or peripheral. The lack of diagnosis in cases of chronic and neuropathic pain in patients with SCD is common, implying inappropriate use of therapeutic resources by the health services, resulting in increased suffering to the patient. The release of inflammatory mediators is related to the perception of pain, and may cause nociceptor sensitization.

The tDCS has the potential to change the neuronal membrane resting potential, this effect is dependent on the polarity, being that cathode produces hyperpolarization, whereas anode produces depolarization, in this way can induce an effect of inhibition and facilitation of neuronal firing, respectively. This effects can induces changes in cortical excitability. Although tDCS may modulate areas related to endogenous pain control, its effects seem to be diffuse, and focality would probably enhance its effects. The peripheral electrical stimulation (PES), in another way, may also modulate cortical excitability, depending mainly on its amplitude and frequency. PES modulation of cortical excitability is very focal, occurring only in the stimulated region. The combination of these two neuromodulatory techniques has showed additive effects in some studies with individuals suffering from chronic pain,which promoting a general effect (tDCS), and the other a more focal effect (TENS). Although this additive effect has been demonstrated, to date, no study evaluate its safety and efficacy in individuals with DF.

As a secondary outcome, the investigators are going to access the influence of the intervention on quantitative electroencephalography (qEEG). Growing evidence points out to different brain characteristics between individuals with chronic pain and healthy. qEEG has high temporal resolution and evaluates primary electrical effects of neural excitation, allowing identify possible patterns of brain functioning in individuals with chronic pain. qEEG allowed the identification of the thalamocortical dysrhythmia (TCD) in patients with chronic pain characterized by an increased low frequency band power density theta (4 - 7Hz) and a decrease in high frequency bands alpha (8 -12Hz) and beta (13 - 30Hz). This dysrhythmic mechanism may occur from the periphery to the thalamus (bottom-up) or cortical dysregulation (top-down), disinhibition of the thalamus. This process results in hyperpolarization of thalamic neurons, leading to a preponderance of low frequency oscillations in qEEG. The persistence thalamic firing at low frequencies can lead to a collateral inhibition in cortical regions around, which could theoretically lead to a decrease in the higher frequencies. This increase occurs at low frequency regions involved in neuro matrix of pain.

The investigators will alse avaluate the influence of the chronic pain sencondary to avascular necrosis of hip joint about cortical motor reorganization using transcranial magnetic stimuation (TMS). Recent data point to a gluteus maximus muscle weakness during maximal voluntary contraction in pronation position in individuals with joint pain in the hip. Similarly, individuals with legg calve perthes who suffer from femoral head necrosis, weakness of the abductor hip musculature was related to poor clinical outcomes. A possible explanation for these findings is cortical motor reorganization, which is associated with motor control impairment, and this has been demonstrated in individuals with chronic lateral epicondylalgia and knee osteoarthritis, where cortical organization is altered and correlated positively with the time of Pain and is associated with the perpetuation of pain. This cortical reorganization can occur in the somatotopic areas corresponding to the motor or sensorial homunculus, having as characteristic an overlap, retraction and "blurring" in the somatotopic representation of a certain region.

The mediators released by cells of the immune and inflammatory system can act directly on neurons sensitizing and enabling them (usually peripheral nociceptors or neurons in the dorsal horn of the spinal cord). There are several mediators in a long and growing list that includes cytokines and neurotrophins.The major cytokines in an acute inflammation are the Tumor Necrosis Factor (TNF) and the interleukins (IL-1), IL-6 and IL-8, which are important mediators of acute and chronic inflammatory reactions, as well as processes of repair and resolution. High serum levels of IL-8 have been observed in patients in vase-occlusive crisis, important clinical aspect of the pathogenesis of SCD. The presence of the mutant allele A appears to influence the expression of the TNF-alpha, being the AA genotype considered a high producer.

Neurotrophins are dimeric proteins that are essential for the normal development of the nervous system in vertebrates. This family includes the nerve growth factor (NGF), brain-derived neurotrophic factor (BDNF) and other neurotrophins (NT). Currently, it is recognized that certain neurotrophins, particularly the NGF and the brain-derived neurotrophic factor BDNF play a significant role in nociception, so that the NGF sensitizes nociceptors at the periphery, while the BDNF enhances the response ability of the dorsal horn neurons of the spinal cord. The BDNF gene, which encodes the BDNF protein, located on chromosome 11 at the boundary of regions 11p13 and 11p14 of the human genome has been investigated in a wide range of areas related to neuroplasticity, including differences in brain morphology, learning and memory, interactions with brain stimulation protocols of plasticity induction and recovery after brain injury and has been associated with a wide variety of neurological disorders, including, for example, depression, schizophrenia and attention deficit hyperactivity disorder (ADHD).

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with sickle cell disease hemoglobin electrophoresis.
* Be aged 18 years old to 50 years old.
* Having signed the consent form and clarified.
* Having chronic pain with at least 3 months duration.
* Being diagnosed with femoral head osteonecrosis
* Have more than one type of chronic pain.

Exclusion Criteria:

* Have cochlear implants, pacemakers or metallic implant in the skull / brain;
* Have metallic implant application site of peripheral stimulation;
* History of head trauma;
* Pregnancy;
* seizures or epilepsy History;
* Being in drug use that modify neuronal activation threshold (eg antidepressants and anticonvulsants);
* Having diagnosis of fibromyalgia, or any impairment to be confused with the symptoms of SCD;
* Have pain confirmed neuropathic type.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-03; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity | One day
  Pain assessment at before and after each intervention:
  Actual pain intensity will be assessed using a 0-10 visual analogue scale (VAS), where 0 is no pain and 10 the worst imaginable pain. Visual analogue scale allows to evaluate the intensity pain of a quantitative way, the subjects will fill a VAS before and after treatment.

SECONDARY OUTCOMES:
Analysis of brain waves delta, theta, alpha and beta | One day
  - Analysis of brain waves: Individuals will be submitted to electroencephalogram following the international classification 10/20 for placement of the electrodes. The researchers will use 30 electrodes referenced by Cz point, ground electrode in Fz point of each individual and the impedance kept below 5 K ohms in all electrodes with a sampling frequency of 600 Hz. All records will be made with closed eyes lasting 4 minutes.
Dosages of TNF-alpha and BDNF in patients with SCD | One day
  - Assessment Dosages of tumor necrosis factor alpha (TNF-alpha) will be properly processed and the serum stored at -20ºC. Detection and quantification of serum levels will be performed by Enzyme-linked Immunosorbent Assay (ELISA) according to the manufacturer's instructions, being considered as normal reference values ≤15 pg / ml for IL-8 and p ≤7,8 / mL for TNF-alpha.
  Dosages of neurotrophin brain-derived neurotrophic factor (BDNF) will be properly processed and the serum stored at -20ºC. The detection and quantification of serum levels will be performed by Enzyme-linked Immunosorbent Assay (ELISA) according to the manufacturer's instructions. The detection limits for the BDNF will be 15 pg/ml.
Motor cortical reorganization | One day
  This outcome will be evaluated with a transcranial magnetic stimulator of single pulse . The procedure consists of ten pulses around the skull vertice with 200μV amplitude.
Impact of pain in functionality | One day
  Assessment of impact of pain in functionality before treatment with a pain disability index (PDI) will be used only in baseline PDI is a 7 questions questionnarie that will be used assess limitations imposed by the presence of pain in daily life activities
Hospital anxiety and depression scale (HADS) | One day
  This scale allows to evaluate objectively both aspects of anxiety and depression. Consists of 2 subscales, each one with 7 items. It will be used to identify the level of anxiety and depression

CONTACTS AND LOCATIONS:
Overall Officials: Abrahão F Baptista, Prof., Principal Investigator — Federal University of Bahia; Wellington S Silva, Prof., Study Director — Faculdade Adventista da Bahia
Locations (1):
- Functional Electrical Stimulation Laboratory, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yusuf HR, Atrash HK, Grosse SD, Parker CS, Grant AM. Emergency department visits made by patients with sickle cell disease: a descriptive study, 1999-2007. Am J Prev Med. 2010 Apr;38(4 Suppl):S536-41. doi: 10.1016/j.amepre.2010.01.001. PMID 20331955
- [Background] Ballas SK. Pain management of sickle cell disease. Hematol Oncol Clin North Am. 2005 Oct;19(5):785-802, v. doi: 10.1016/j.hoc.2005.07.008. PMID 16214644
- [Background] Lima MC, Riberto M, Batistella LR, Boggio PS, Fregni F. Estimulação cerebral para o tratamento de dor neuropática. Psicol. teor. prát. 2007; 9(2):142-149
- [Background] Oliveira LB, Lopes TS, Soares C, Maluf R, Goes BT, Sa KN, Baptista AF. Transcranial direct current stimulation and exercises for treatment of chronic temporomandibular disorders: a blind randomised-controlled trial. J Oral Rehabil. 2015 Oct;42(10):723-32. doi: 10.1111/joor.12300. Epub 2015 Apr 20. PMID 25891021
- [Background] Brunoni AR, Pinheiro FS, Boggio PS. Estimulação transcraniana por corrente contínua: in Fregni F, Boggio PS, Brunoni AR. Neuromodulação Terapêutica: Princípios e Avanços da Estimulação cerebral não invasiva em Neurologia, reabilitação, Psiquiatria e Neuropsicologia. São Paulo: Sarvier. 2012: 65-75.
- [Background] Boggio PS, Amancio EJ, Correa CF, Cecilio S, Valasek C, Bajwa Z, Freedman SD, Pascual-Leone A, Edwards DJ, Fregni F. Transcranial DC stimulation coupled with TENS for the treatment of chronic pain: a preliminary study. Clin J Pain. 2009 Oct;25(8):691-5. doi: 10.1097/AJP.0b013e3181af1414. PMID 19920718
- [Background] Schabrun SM, Jones E, Elgueta Cancino EL, Hodges PW. Targeting chronic recurrent low back pain from the top-down and the bottom-up: a combined transcranial direct current stimulation and peripheral electrical stimulation intervention. Brain Stimul. 2014 May-Jun;7(3):451-9. doi: 10.1016/j.brs.2014.01.058. Epub 2014 Jan 30. PMID 24582372
- [Background] Hazime FA, de Freitas DG, Monteiro RL, Maretto RL, Carvalho NA, Hasue RH, Joao SM. Analgesic efficacy of cerebral and peripheral electrical stimulation in chronic nonspecific low back pain: a randomized, double-blind, factorial clinical trial. BMC Musculoskelet Disord. 2015 Jan 31;16(1):7. doi: 10.1186/s12891-015-0461-1. PMID 25636503
- [Background] Vuckovic A, Hasan MA, Fraser M, Conway BA, Nasseroleslami B, Allan DB. Dynamic oscillatory signatures of central neuropathic pain in spinal cord injury. J Pain. 2014 Jun;15(6):645-55. doi: 10.1016/j.jpain.2014.02.005. Epub 2014 Mar 1. PMID 24589821
- [Background] de Vries M, Wilder-Smith OH, Jongsma ML, van den Broeke EN, Arns M, van Goor H, van Rijn CM. Altered resting state EEG in chronic pancreatitis patients: toward a marker for chronic pain. J Pain Res. 2013 Nov 25;6:815-24. doi: 10.2147/JPR.S50919. PMID 24379694
- [Background] Sarnthein J, Stern J, Aufenberg C, Rousson V, Jeanmonod D. Increased EEG power and slowed dominant frequency in patients with neurogenic pain. Brain. 2006 Jan;129(Pt 1):55-64. doi: 10.1093/brain/awh631. Epub 2005 Sep 23. PMID 16183660
- [Background] Apkarian AV, Bushnell MC, Treede RD, Zubieta JK. Human brain mechanisms of pain perception and regulation in health and disease. Eur J Pain. 2005 Aug;9(4):463-84. doi: 10.1016/j.ejpain.2004.11.001. Epub 2005 Jan 21. PMID 15979027
- [Background] Michels L, Moazami-Goudarzi M, Jeanmonod D. Correlations between EEG and clinical outcome in chronic neuropathic pain: surgical effects and treatment resistance. Brain Imaging Behav. 2011 Dec;5(4):329-48. doi: 10.1007/s11682-011-9135-2. PMID 21948245
- [Background] Boord P, Siddall PJ, Tran Y, Herbert D, Middleton J, Craig A. Electroencephalographic slowing and reduced reactivity in neuropathic pain following spinal cord injury. Spinal Cord. 2008 Feb;46(2):118-23. doi: 10.1038/sj.sc.3102077. Epub 2007 May 15. PMID 17502876
- [Background] Llinas RR, Ribary U, Jeanmonod D, Kronberg E, Mitra PP. Thalamocortical dysrhythmia: A neurological and neuropsychiatric syndrome characterized by magnetoencephalography. Proc Natl Acad Sci U S A. 1999 Dec 21;96(26):15222-7. doi: 10.1073/pnas.96.26.15222. PMID 10611366
- [Background] Goncalves MS, Queiroz IL, Cardoso SA, Zanetti A, Strapazoni AC, Adorno E, Albuquerque A, Sant'Ana A, dos Reis MG, Barral A, Barral Netto M. Interleukin 8 as a vaso-occlusive marker in Brazilian patients with sickle cell disease. Braz J Med Biol Res. 2001 Oct;34(10):1309-13. doi: 10.1590/s0100-879x2001001000011. PMID 11593306
- [Background] Hajeer AH, Hutchinson IV. Influence of TNFalpha gene polymorphisms on TNFalpha production and disease. Hum Immunol. 2001 Nov;62(11):1191-9. doi: 10.1016/s0198-8859(01)00322-6. PMID 11704281
- [Background] Louis E, Franchimont D, Piron A, Gevaert Y, Schaaf-Lafontaine N, Roland S, Mahieu P, Malaise M, De Groote D, Louis R, Belaiche J. Tumour necrosis factor (TNF) gene polymorphism influences TNF-alpha production in lipopolysaccharide (LPS)-stimulated whole blood cell culture in healthy humans. Clin Exp Immunol. 1998 Sep;113(3):401-6. doi: 10.1046/j.1365-2249.1998.00662.x. PMID 9737669
- [Background] Moalem G, Tracey DJ. Immune and inflammatory mechanisms in neuropathic pain. Brain Res Rev. 2006 Aug;51(2):240-64. doi: 10.1016/j.brainresrev.2005.11.004. Epub 2006 Jan 4. PMID 16388853
- [Background] Chaieb L, Antal A, Ambrus GG, Paulus W. Brain-derived neurotrophic factor: its impact upon neuroplasticity and neuroplasticity inducing transcranial brain stimulation protocols. Neurogenetics. 2014 Mar;15(1):1-11. doi: 10.1007/s10048-014-0393-1. Epub 2014 Feb 25. PMID 24567226